CLINICAL TRIAL: NCT00083941
Title: Clinical Trial Phase II (Single Centre Study) : A Preliminary Study of the Safety, Immunogenicity, and Clinical Efficacy of TroVax Given in Conjunction With Interleukin 2 (IL-2) in the Treatment of Stage IV Renal Cell Cancer
Brief Title: A Study of TroVax Vaccine Given in Conjunction With IL-2 for Treatment of Stage IV Renal Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oxford BioMedica (Industry)
Collaborators: Columbia University (Other); ORION Clinical Services (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TV2 Renal
Record Dates: First submitted 2004-06-03; First posted 2004-06-07 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Carcinoma, Renal Cell
Keywords: Renal Cell Cancer; Requiring IL-2 treatment; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — TroVax; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TroVax and IL-2 (Experimental): TroVax: Intramuscular into the deltoid muscle of the upper arm, 10x dose (6.83 x 108 pfu/ml). IL 2: High dose IL 2, 600,000 IU/kg intravenously every 8 hours up to a maximum of 15 injections.
  Interventions: Biological: TroVax; Biological: Interleukin-2

INTERVENTIONS:
Biological: TroVax — 1ml intramuscular injection
Biological: Interleukin-2 — Intravenous IL-2
  Other Names: IL-2

SUMMARY:
The purpose of this study is to test the safety of an investigational vaccine called TroVax when given in conjunction with Interleukin-2 (IL-2) treatment. TroVax is the experimental product in this trial and its value as a medicine has not yet been proven. Interleukin-2 (IL-2) is standard treatment for your cancer, which means that you could receive it even if you choose not to participate in this study. TroVax is being studied as a possible treatment for patients with cancer of the kidney.

TroVax belongs to a class of medicines called a vaccine. A vaccine helps the body's immune system to recognize and kill foreign invading organisms effectively. It is believed that one of the reasons why cancer can spread through the body is that the immune system cannot recognize them as being different from normal tissues and therefore cannot kill the cancer cells. A vaccine that alerts the immune system to the presence of cancer cells in the body could lead to the immune system being able to target and kill those cancer cells effectively. This trial is of a completely new way of trying to treat cancer in the future by the use of vaccination injections. TroVax consists of a virus that has been changed so that it is no longer infectious and carries a gene for a protein called 5T4. This protein is carried by many kidney cancer calls. When the virus is injected, it makes the protein, and the body's immune system is then able to recognize this protein and kill the cells that have it (i.e. the cancer cells).

The purpose of this study is to assess the safety and tolerability of TroVax injections and to understand whether TroVax could make such an immune response happen in patients with renal cell cancer while receiving Interleukin-2 (IL-2). This study will also observe and monitor any side effects experienced in patients who receive TroVax while being treated with IL-2.

DETAILED DESCRIPTION:
Objectives

Primary

* To assess the safety and tolerability of TroVax injections when given as a therapeutic vaccine to patients with metastatic renal cell cancer
* To assess the immune responses induced by treatment with TroVax

Secondary

* To assess the impact of treatment with TroVax on tumour response rates, time to disease progression and two year survival.

Study design This will be an open label evaluation of the combination of TroVax with IL-2. The dosage regimen will be injections of TroVax given at three weekly intervals commencing before treatment with IL-2 (one treatment) and then in conjunction with IL-2 for up to four treatments. Following completion of treatment with IL-2, booster injections of TroVax will be given at three monthly intervals for a further three injections to patients whose disease responds or stabilises after treatment with IL-2 and TroVax.

The first dose of TroVax will be given alone to allow an initial safety assessment. The second dose will be given with the standard institutional regimen of high dose IL-2. IL-2 will be given for 5 consecutive days every three weeks for two or more (typically four) cycles provided that the patients are responding to treatment (i.e. tumour response or stabilisation). The first dose of IL-2 will be given starting on the same day as the second TroVax injection. If the patient does not tolerate treatment with IL-2, dosing with TroVax will continue on a three weekly cycle until a total of 5 injections has been given (week 12). Following this, TroVax boosters will be given every at six, nine and 12 months providing that the disease remains stable or responding. The total treatment period may last for up to 12 months with a further follow up period of up to 12 months (total study period 24 months).

All patients will be followed up to assess tolerability, induction of humoural and cellular immunity to 5T4 cell surface antigen and immune response to the vector. The tumour will be restaged after every two cycles of IL-2 treatment by CT scans, in accordance with current institutional and clinical guidelines. Once treatment with IL-2 has stopped, boosting and restaging will occur every 3 months for a total treatment period of up to one year. Once this treatment has stopped, patients will be followed for a further twelve months, with CT scans every 3 months (standard of care). If at the end of that period, the patient still has stable or responding disease, that patient will be followed at three monthly intervals until disease progression occurs.

If the patients' disease progresses at any stage or serious or severe adverse drug reactions relating to TroVax occur, treatment with TroVax will cease but patients should be kept on study and followed three monthly until they have been on study for 24 months. Other treatments for the cancer will be recorded in the CRF.

A total of 25 patients will be enrolled.

Study population Inclusion criteria

1. Metastatic renal clear cell adenocarcinoma, histologically proven by biopsy of the primary tumour and/or a metastasis. If a fresh specimen is obtained for diagnostic purposes, it may be frozen and stained for 5T4. Prior nephrectomy is not required.
2. Requiring treatment with IL-2 and able to tolerate a high dose schedule per institutional standards.
3. Aged 18 years or more.
4. Performance status (ECOG) 0 or 1.
5. Expected survival longer than three months.
6. No clinically active autoimmune disease.
7. Total white cell count ≥ 3 x 109/l.
8. Platelet count ≥ 90,000/mm3.
9. Serum creatinine 1.6 mg/dl or less.
10. Total bilirubin 1.6 mg/dl or less.
11. Serum AST/ALT ≥ three times the upper limit of normal or 5 times upper limit of normal if liver metastases are present.
12. Able to give written informed consent and to comply with the protocol.
13. Women must be either post menopausal, rendered surgically sterile or practising a reliable form of contraception (hormonal, intrauterine device or barrier). Men must practise an effective form of birth control, such as barrier protection.
14. Normal cardiac stress test if the patients are older than 50 years of age or have symptoms of cardiac disease.
15. Normal pulmonary function tests if the patient is a smoker or is known to have primary lung disease.

Exclusion criteria

1. Pregnancy, lactation or lack of effective contraception in fertile men and women of childbearing potential.
2. Intercurrent serious infections within the 28 days prior to entry to the trial.
3. Known to be HIV positive because HIV infection can lead to serious adverse events with vaccination and/or high-dose IL-2.
4. Life threatening illness unrelated to cancer.
5. Cerebral metastases.
6. History of allergic response to previous vaccinia vaccinations.
7. Participation in any other clinical trial within the previous 30 days .
8. Previous malignancies within the last two years other than successfully treated squamous carcinoma of the skin or in situ carcinoma of the cervix treated with cone biopsy.
9. Previous history of major psychiatric disorder requiring hospitalisation or any current psychiatric disorder that would impede the patient's ability to provide informed consent or to comply with the protocol.
10. Corticosteroids unless used as an antiemetic.
11. Family contact with active eczema, exfoliative skin disorder, pregnancy or other cause of immunocompromise.

Withdrawal criteria

1. Non-compliance with the protocol.
2. Patient request.
3. Physician decision.
4. Concurrent involvement in a clinical trial of any other drug. Treatment plan and methods This will be an open label evaluation of the combination of TroVax with IL-2. The dosage regimen will be three injections of TroVax given every three weeks. The first vaccine will be given alone. The second and third vaccine will be given at weeks 3 and 6 with IL-2 commencing immediately after vaccination. If there is no evidence of disease progression on the week 9 CT scans (chest, abdomen, pelvis), an additional two cycles of TroVax and IL-2 will be given at weeks 9 and 12. Following completion of treatment with IL-2, booster injections of TroVax will be given at three monthly intervals for a further three injections, provided patients have stable or responding disease.

Patients complying with the entry criteria will be invited to enter the study. After giving fully informed consent, patients will be subjected to a medical history and physical examination to document general fitness to proceed with the trial. Previous exposure to small pox vaccine will be noted. The diagnosis should be confirmed histologically from the patient's records. If possible, a retained sample will be obtained to stain for 5T4. If a fresh sample is taken, it may be cryopreserved and also examined for 5T4. At that time, metastases will be documented using relevant CT scans (chest, abdomen, pelvic). An MRI scan of the brain will be obtained. A cardiac stress test and pulmonary function tests will be obtained in appropriate patients.

Blood will also be drawn for haematology and clinical chemistry, full blood count with differential white cell and platelet counts, urea and electrolytes, liver function tests (total bilirubin, AST, ALT, GGT, alkaline phosphatase), serum proteins, calcium, phosphate, glucose and creatinine), pituitary hormone screen (ACTH, TSH, LH, FSH;), antinuclear and anti-skeletal muscle antibodies and immunological testing (antibodies to 5T4 and vector, cellular responses to 5T4; 100 ml). In potentially fertile women, a pregnancy test will be obtained. A urine sample will be obtained for urinalysis for protein and blood. This screen should not occur more than two weeks before the immunisation schedule begins.

At week 0, the patients will be immunised with a single intramuscular injection of 1 ml of TroVax 10x. This dose will be given without IL-2. Then, every three to four weeks for four injections, TroVax will be given in the morning. These doses may be given in conjunction with IL-2. Immediately before each injection, blood will be drawn for immunological testing (100 ml). Before the injection, blood will also be drawn for clinical pathology (full blood count and clinical chemistry). A urine sample will be obtained for urinalysis for protein and blood.

IL-2 will be given intravenously (IV) in a dose of 600,000 IU/kg every eight hours for up to 15 injections in each cycle. The first dose will be given in the afternoon of the same day as the second TroVax injection. These cycles of TroVax and IL-2 will be repeated every 3-4 weeks depending upon patient tolerance and clinical response. Cycles of IL-2 will always commence in the afternoon after TroVax has been given in the morning. If IL-2 is not tolerated, it may be suspended but treatment with TroVax will be continued so long as it is well tolerated. TroVax may be given for up to three months (i.e. injection 5) to patients with progressive disease so long as no other anticancer treatment (i.e. chemotherapy, interferon alpha or radiotherapy) is considered indicated for them.

CT scans (chest abdomen, pelvis) will be obtained to restage the disease at weeks 9-10 and 15-16 (i.e. after two and four doses of IL-2 and/or 3 and 5 doses of TroVax).

A blood sample for immunological testing (100 ml) will be obtained three and eight weeks after the fifth TroVax injection (4 and 5 months).

Following the CT scan at 15-16 weeks patients will be followed at three monthly intervals, commencing at six months. Patients whose disease is progressing at this point may not be treated further with TroVax but may be kept on study and observed at three monthly intervals. Patients whose disease has stabilised or responded will be offered three further injections of TroVax at months 6, 9 and 12. Patients whose disease progresses or who experience serious or severe adverse events related to TroVax will stop treatment with TroVax but may be kept on study and reviewed at three monthly intervals. If the patient requires further treatment with established anticancer agents, these will be recorded in the CRF.

At each visit, from week 12 to month 12, regardless of disease status, blood will be obtained (prior to the injection of TroVax, if indicated) for clinical pathology, pituitary hormone screen, autoantibodies and immunological testing (100 ml). A urine sample will be obtained for urinalysis for protein and blood. The disease will be restaged using CT scans (chest abdomen, pelvis).

When TroVax is being administered, patients will return 3 weeks after each TroVax injection for immunological testing (100 ml).

After month 12, patients will return at three monthly intervals for a further 12 months. At each visit, the disease will be restaged using CT scans (chest abdomen, pelvis) in accordance with current institutional guidelines. Blood (100 ml) will be obtained for immunological testing, autoantibodies and pituitary function tests. A urine sample will be obtained for urinalysis for protein and blood. Patients, who at the end of this period, have stable or responding disease may be followed at three monthly intervals until disease progression occurs.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic renal clear cell adenocarcinoma, histologically proven by biopsy of the primary tumour and/or a metastasis. If a fresh specimen is obtained for diagnostic purposes, it may be frozen and stained for 5T4. Prior nephrectomy is not required.
* Requiring treatment with IL-2 and able to tolerate a high dose schedule per institutional standards.
* Aged 18 years or more.
* Performance status (ECOG) 0 or 1.
* Expected survival longer than three months.
* No clinically active autoimmune disease.
* Total white cell count greater than or equal to 3 x 109/l.
* Platelet count greater than or equal to 90,000/mm3.
* Serum creatinine 1.6 mg/dl or less.
* Total bilirubin 1.6 mg/dl or less.
* Serum AST/ALT greater than or equal to three times the upper limit of normal or 5 times upper limit of normal if liver metastases are present.
* Able to give written informed consent and to comply with the protocol.
* Women must be either post menopausal, rendered surgically sterile or practising a reliable form of contraception (hormonal, intrauterine device or barrier). Men must practise an effective form of birth control, such as barrier protection.
* Normal cardiac stress test if the patients are older than 50 years of age or have symptoms of cardiac disease.
* Normal pulmonary function tests if the patient is a smoker or is known to have primary lung disease.

Exclusion Criteria:

* Pregnancy, lactation or lack of effective contraception in fertile men and women of childbearing potential.
* Intercurrent serious infections within the 28 days prior to entry to the trial.
* Known to be HIV positive because HIV infection can lead to serious adverse events with vaccination and/or high-dose IL-2.
* Life threatening illness unrelated to cancer.
* Cerebral metastases.
* History of allergic response to previous vaccinia vaccinations.
* Participation in any other clinical trial within the previous 30 days .
* Previous malignancies within the last two years other than successfully treated squamous carcinoma of the skin or in situ carcinoma of the cervix treated with cone biopsy.
* Previous history of major psychiatric disorder requiring hospitalisation or any current psychiatric disorder that would impede the patient's ability to provide informed consent or to comply with the protocol.
* Corticosteroids unless used as an antiemetic.
* Family contact with active eczema, exfoliative skin disorder, pregnancy or other cause of immunocompromise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2004-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
To assess safety and tolerability of TroVax | duration of study
  incidence of adverse events, laboratory tests and occurrence of dose limiting toxicity
To assess immune responses induced by treatment with TroVax | duration of study
  positive antibody response for the vector (MVA) / tumour (5T4)

CONTACTS AND LOCATIONS:
Overall Officials: Howard L Kaufman, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia Presbyterian Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kaufman HL, Taback B, Sherman W, Kim DW, Shingler WH, Moroziewicz D, DeRaffele G, Mitcham J, Carroll MW, Harrop R, Naylor S, Kim-Schulze S. Phase II trial of Modified Vaccinia Ankara (MVA) virus expressing 5T4 and high dose Interleukin-2 (IL-2) in patients with metastatic renal cell carcinoma. J Transl Med. 2009 Jan 7;7:2. doi: 10.1186/1479-5876-7-2. PMID 19128501